CLINICAL TRIAL: NCT01329302
Title: Follicular Flushing for Poor Responder Patient in an Assisted Reproductive Technology Program: Flush Study
Brief Title: Benefit of Follicular Flushing During Oocyte Retrieval for Poor Responder Patient in an Assisted Reproductive Technology Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2010-A00589-30
Record Dates: First submitted 2010-12-22; First posted 2011-04-05 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Infertility, Female; Ovarian Insufficiency
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Direct aspiration (Active Comparator)
  Interventions: Procedure: Direct aspiration needle Echo tip® Cook® single Lumen and Follicular flushing with double lumen needle Echo tip® Cook® Double Lumen Aspiration
- Follicular Flushing (Active Comparator)
  Interventions: Procedure: Direct aspiration needle Echo tip® Cook® single Lumen and Follicular flushing with double lumen needle Echo tip® Cook® Double Lumen Aspiration

INTERVENTIONS:
Procedure: Direct aspiration needle Echo tip® Cook® single Lumen and Follicular flushing with double lumen needle Echo tip® Cook® Double Lumen Aspiration — In addition to direct aspiration of the follicular fluid all follicles are flushed with flushing solution, 20CC of flushing medium( Flushing Medium MediCultâ France) is provided for all the procedure and flushing medium is collected separately from direct fluid

SUMMARY:
The object of this study is to determine the benefit of follicular flushing with a double channel needle in a poor responder population for a maximum number of oocytes to be retrieved. The investigators compare two methods of oocyte retrieval with or without flushing. 220 patients undergoing an in vitro fertilization (IVF) or Intracytoplasmic Sperm Injection (ICSI) have to be included. All patients with less than 5 follicles of 14 mm and more the day of ovulation induction will be included, following a randomized protocol in two groups, Group A: Oocyte retrieval is performed with a single lumen aspiration needle 17G. Group B: Oocyte retrieval is performed with a double lumen aspiration needle 17G. all follicles are flushed with flushing solution in addition to direct aspiration of the follicular fluid, 20CC of flushing medium is provided for all the procedure and flushing medium is collected separately from direct fluid aspiration in order to follow up each oocyte one by one. First criterion of our comparison is the number of oocyte retrieved. Second criteria are: oocyte quality, fertilization rate, number and quality of embryos obtained, clinical pregnancy rate. In Group B the investigators will compare two subgroups: oocytes collected in flush medium and oocytes from direct follicle fluid. Then the investigators will know the capability of oocyte collected after follicular flushing to be fertilized and to increase the success chance of pregnancy for poor responder patients.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing an IVF or ICSI treatment
* long agonist, antagonist or short stimulations protocols
* less than 5 follicles of 14mm or more day of HCG
* Major patients aged under 43 years
* patient within a couple married or can prove a married life of over 2 years

Exclusion Criteria:

* all the cons indication to the oocyte retrieval
* oocyte donor
* Couple supported viral loop
* Patient does not speak French or unable to give informed consent
* Patients major protected
* Patients with biopsy performed on weekends are also excluded due to unavailability of adequate personnel and equipment
* Absence of follicles

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
the number of mature oocytes collected | 2 years and 9 months
  Increase the number of mature oocytes collected during the follicular flushing with a double lumen aspiration needle
quality of embryos obtained | 2 years and 9 months
  Embryo quality is assessed at the Laboratory of Reproductive Biology by a score based on: cell number, cell regularity and degree of fragmentation.

SECONDARY OUTCOMES:
Number of embryos obtained | 2 years and 9 months
Number of transferable embryos (transferred and frozen) | 2 years and 9 months
  Biologist at Day 3 chooses the best quality embryos for transfer and freeze the other if the quality is sufficient.
Number of pregnancies obtained | 2 years and 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Assistance Médicale à la Procréation, CMCO-SIHCUS, Schiltigheim, Schiltigheim, France

REFERENCES:
- [Result] Calabre C, Schuller E, Goltzene MA, Rongieres C, Celebi C, Meyer N, Teletin M, Pirrello O. Follicular flushing versus direct aspiration in poor responder IVF patients: a randomized prospective study. Eur J Obstet Gynecol Reprod Biol. 2020 May;248:118-122. doi: 10.1016/j.ejogrb.2020.03.003. Epub 2020 Mar 6. PMID 32200248